CLINICAL TRIAL: NCT03182283
Title: Person-Centered Psychosis Care: An Educational Intervention for Inpatient Staff
Brief Title: Person-Centered Psychosis Care: An Educational Intervention
Acronym: PCPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: PCPC
Record Dates: First submitted 2017-05-17; First posted 2017-06-09 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Patient-Centered Care; Psychiatry; Inpatient; Psychosis
Keywords: Person-centered care; Psychosis care; Integrated care
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Non-randomized before and after design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): All patients at the psychosis wards receive care as usual before staff goes through educational intervention.
- Post-intervention (Other): After staff attended educational intervention and implemented Person-centered psychosis care in the wards all patients admitted will receive person-centered care.
  Interventions: Behavioral: Person-centered psychosis care

INTERVENTIONS:
Behavioral: Person-centered psychosis care — Person-centered care educational intervention for staff with following implementation of person-centered care in the clinic
  Arms: Post-intervention

SUMMARY:
Schizophrenia is a major mental illness that presents in young adulthood and affects ~1% of the population. Impact on affected persons life is often major and life expectancy is reduced by ~20 years. Better and more effective care models are needed to increase health in these persons. Person-centered care have been suggested to be one way to increase efficiency in care delivery for patients with chronical and complex conditions. The impact of person-centered care on a inpatient psychosis care setting is now being tested.

The purpose of this study is to test whether inpatient Person-centered psychosis care (PCPC) can

1. increase patient empowerment
2. improve patient satisfaction
3. reduce the frequency of involuntary treatments
4. reduce the duration of inpatient care and
5. reduce overall ward burden

A further purpose is to qualitatively explore which components in this complex intervention are experienced as facilitators or barriers to the achievement of good care, from both patient, next-of-kin and staff perspectives.

Quantitative data is collected through questionnaires from patients (measuring empowerment, care satisfaction and perceived health) before and after an educational intervention for staff, along with ward level measures such as care burden, number of involuntary treatments and length of stay on ward.

Qualitative interview is used to study experiences of patients, next-of-kin and staff.

DETAILED DESCRIPTION:
Background

Schizophrenia is a major mental illness that presents in young adulthood. It affects approximately 1% of the population and is a major cause of Disability-adjusted Life Years worldwide. Besides impacting on the ability to independently carry out daily activities, work/studies and interactions with family and community, the illness has a profound effect on physical health. Diabetes and cardiovascular diseases are common complications and life expectancy is reduced by as much as two decades. The long term nature of this complex illness highlights the need for more effective, holistic care models. Increased patient involvement is central, as it has been shown that patients' views of appropriate interventions often differ from those of formal care providers.

Person-centered care (PCC) is recognized by the WHO as a valuable approach to the care of chronic conditions. A basic assumption of person-centered care (PCC) is that healthcare must recognize the patient as a person, with own knowledge, capacity and preferences along with needs and problems. The PCC way to deal with illness and disease is to form a partnership with the person and together form a plan of action to increase health (i.e. not only focus on symptoms or signs of diagnosed disease) taking into account the person's context and priorities. Previous studies show that persons with serious mental illness can and want to participate in their own care and participation might increase adherence. Improved social function and consumer satisfaction were demonstrated when a person-centered care approach, Integrated Care (IC) was tested in a psychosis outpatient-based randomized controlled trial.

To the best of the authors knowledge, PCC has yet to be tested in an inpatient setting for persons with severe mental illness. Favorable results have been demonstrated with regard to both ward level and patient level outcomes from inpatient settings within somatic care. Person-centered care in geriatric settings, which might share some common issues with hospital care for persons with schizophrenia (decreased cognitive function, lack of insight, compromised autonomy), have shown positive outcomes for QoL and agitation in patients and job satisfaction for staff. Reviews show mixed results though. Thus, we wanted to evaluate an intervention for inpatient psychiatric care for persons with schizophrenia and similar psychoses. To this end, we developed Person-centered Psychosis Care (PCPC), a staff educational intervention involving components of PCC as well as IC. Person Centered Psychosis Care was defined as having four key elements; dialogue, building partnership, formulation and documentation of a health plan, and early involvement of the patient's outpatient facility. The latter means that the patient's outpatient-based social resource group can come into play already during the inpatient stay.

Purpose

The purpose of this study is to test whether inpatient PCPC can

1. increase patient empowerment
2. improve patient satisfaction
3. reduce the frequency of involuntary treatments
4. reduce the duration of inpatient care and
5. reduce overall ward burden

   A further purpose is to qualitatively explore which components in this complex intervention are experienced as facilitators or barriers to the achievement of good care, from both patient, next-of-kin and staff perspectives.

   Methods

   The study employs a simple "before and after" design. Quantitative data (patient-level, ward-level) are collected pre- and post intervention on all four wards. Qualitative data are provided through interviews with patients as well as focus groups with staff.

   Data collection: Patient-level data All patients on any of the four wards who fulfill study criteria during pre- and post-intervention periods will be asked to participate in the study.

   Anticipated number of participants: 50 pre intervention, 50 post intervention.Those who accept will complete questionnaires at the clinic together with the interviewer. The following outcomes will be measured:
   * Empowerment will be measured with The Empowerment Scale. This scale is validated and used internationally in studies involving persons with severe mental ill-health. There are 28 questions; responses are given on a scale of 1 (agree totally) to 4 (disagree totally).
   * Patient satisfaction measured with the UKU-ConSat Rating Scale consists of 11 items on different aspects of the care provided where response is given on a scale 1 (Very bad/negative/little) to 7 (very good/positive/much). The scale also includes two VAS-like scales where an answer is marked on a 100 mm line to a question on overall life experience (0=worst imaginable, 100=best imaginable).

   Confounders including illness burden, functional ability, and overall health will be quantified for each patient at discharge. Positive and negative symptom burden will be rated with the Remission subscale of PANSS, consisting of 8 items reflecting core symptoms of schizophrenia and functional ability will be determined using the GAF scale and overall health with the EQ-5D. Ratings will be carried out by two nurses and one psychologist.

   After the completion of the scales, all participants are asked the following open-ended questions:

   1a) What are the most important things that have improved for you during your stay at the hospital?

   1b) What was the reason that you got better? 2a) What do you wish could improve for you in the future, after your hospital stay? 2b) How could the health care sector help you to achieve this?

   At the end of the interview, participants are asked for permission for researchers to contact them after discharge for invitation to a qualitative interview study. A purposive selection of stabilized patients who accepted follow-up contact will be asked if they would like to participate in an interview with a study nurse or psychologist. The interview will focus on experiences of care during the inpatient stay and patient-relevant endpoints will be explored. The sampling will aim at a heterogeneous group with regard to gender, age, ethnicity, level of psychosocial function, involuntary vs voluntary care.

   Data collection: Next-of-kin A purposive sample of family members or other persons close to the patient will be asked if they would like to participate in focus groups/an interview. The selection of family members' for focus group interview will strive to include next-of-kin of patients with varied backgrounds with regard to age, gender, ethnic background, education level, living situation (do they live together with the patient or not?) etc. The main focus for this focus group will be the identification of positive and negative experiences in the care, discrimination, facilitators and barriers for good care

   Data collection: Staff experiences A purposive sample of staff were invited to participate in focus group to collect experiences of the educational intervention and implementation. Facilitators and barriers to implementation of PCPC will be in focus. Staff were recruited through invitation via e-mail and posters on their wards. In a second step section leaders at the wards asked persons who would be on duty on the days of interview to participate. All focus groups are led by an experienced clinician with research experience of qualitative studies. All interviews will be recorded and transcribed verbatim.

   Data collection: Ward level data Mean number of inpatient days, mean number of inpatient days with compulsory care and mean number of involuntary treatment interventions (involuntary injections, medical restraint) for pre- and post intervention periods will be derived from the clinic's administrative database. Overall care burden is measured at each ward with an instrument developed by the Psychosis Clinic for quality monitoring. The instrument includes objective items (number of admissions and discharges, number of involuntary treatments during the shift etc), followed by a subjective item on the overall level of burden perceived during the shift. The form is filled out by one staff member on each ward once a day according to clinical routine.

   Data analysis: Quantitative data The main study question is whether the intervention is associated with a change in the degree of empowerment experienced by persons who receive hospital care due to psychosis. The secondary outcome measure is patient satisfaction at discharge. Quantitative ratings before and after the care intervention will be compared with standard statistical methods. Similarly, for the ward level analyses, wardwide outcomes will be compared in wards before and after the implementation of the intervention: mean number of inpatient days, mean number of inpatient days with compulsory care, mean number of involuntary treatment interventions and overall ward burden. Distribution of the variables to be studied will determine whether parametric or non-parametric analyses are employed.

   Data analysis: Qualitative data Free text responses to the open-ended questions at the end of the quantitative interview (see patient level data above) as well as data from individual patient interviews and focus group interviews with staff and next-of-kin will be analyzed using content analysis and thematic analysis.

   Ethics All participants (patients, next-of kin and staff) are given written and oral information about the study, the voluntary participation, possibility to withdraw from participation without having to give explanation. All will sign consent form before participating in any study related task, a copy of signed consent is given participants. The study was approved by the Regional Ethics Board in Gothenburg, Dnr. 773-13.

   Time plan Data collection for the pre-intervention phase is completed (December 2014); the educational intervention is completed (May 2015) and the implementation period will end April 30, 2017. Focus group interviews with staff regarding the educational package are now underway (2017). Audit to determine the level of PCPC implementation is currently underway (April 2017), which will determine whether post-intervention data collection could start. Complete data set should be available fall 2017.

   Comment on project so far

   This is a complex intervention involving action research and the study is registered first after the completion of the educational intervention and on-ward implementation of PCPC. The implementation process has been dynamic and varied at the four different wards involved in the project. The duration of the implementation period was considerably longer than anticipated. This is in part related to high staff turnover, serious lack of psychiatrically trained RNs, as well as other barriers to implementation. Barriers have slowly been overcome by changes in routines instigated from within the care staff (as opposed to being imposed on staff from "above"). While the long implementation process can be seen as a limitation, it's interactive nature can at the same time be construed as a strength, as change from within can be expected to increase sustainable change.

   A quantitative study was planned with questionnaires investigating consumer satisfaction and care giver burden in next-of-kin but baseline collection resulted in too few participants to continue that subproject.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psychotic illness in accordance with ICD-10
* Medically ready for discharge as deemed by ward psychiatrist

Exclusion Criteria:

* Severe cognitive disability
* Lack of basic Swedish language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04-25 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in patient empowerment (between before and after cohorts) | Baseline (for before-intervention cohort), 2 years (for after-intervention cohort)
  Patient reported empowerment measured by The Empowerment Scale (Rogers et al 2010).

SECONDARY OUTCOMES:
Change in consumer satisfaction (between before and after cohorts) | Baseline (for before-intervention cohort), 2 years (for after-intervention cohort)
  Patients satisfaction with different aspects of care measured by UKU-ConSat Rating Scale (Ahlfors et al 2000).
Change in staff care burden (before and after intervention and implementation) | Baseline, 2 years
  Overall care burden as reported by staff daily (objective and subjective items) in an internal instrument used by the Psychosis Clinic for quality monitoring.
Change in inpatient days with/out involuntary care (between before and after cohorts) | Baseline (for before-intervention cohort), 2 years (for after-intervention cohort)
  Mean number of inpatient days, mean number of inpatient days with compulsory care.
Change in involuntary treatment (between before and after cohorts) | Baseline (for before-intervention cohort), 2 years (for after-intervention cohort)
  Mean number of involuntary treatment interventions (involuntary injections, medical restraint)

CONTACTS AND LOCATIONS:
Overall Officials: Margda Waern, Professor, Principal Investigator — Göteborg University & Sahlgrenska University Hospital; Anneli Goulding, Phd, Study Director — Sahlgrenska University Hospital & Göteborg University
Locations (1):
- Psychosis Clinic, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossler W, Salize HJ, van Os J, Riecher-Rossler A. Size of burden of schizophrenia and psychotic disorders. Eur Neuropsychopharmacol. 2005 Aug;15(4):399-409. doi: 10.1016/j.euroneuro.2005.04.009. PMID 15925493
- [Background] von Hausswolff-Juhlin Y, Bjartveit M, Lindstrom E, Jones P. Schizophrenia and physical health problems. Acta Psychiatr Scand Suppl. 2009;(438):15-21. doi: 10.1111/j.1600-0447.2008.01309.x. PMID 19132962
- [Background] Tiihonen J, Lonnqvist J, Wahlbeck K, Klaukka T, Niskanen L, Tanskanen A, Haukka J. 11-year follow-up of mortality in patients with schizophrenia: a population-based cohort study (FIN11 study). Lancet. 2009 Aug 22;374(9690):620-7. doi: 10.1016/S0140-6736(09)60742-X. PMID 19595447
- [Background] Lasalvia A, Boggian I, Bonetto C, Saggioro V, Piccione G, Zanoni C, Cristofalo D, Lamonaca D. Multiple perspectives on mental health outcome: needs for care and service satisfaction assessed by staff, patients and family members. Soc Psychiatry Psychiatr Epidemiol. 2012 Jul;47(7):1035-45. doi: 10.1007/s00127-011-0418-0. Epub 2011 Aug 18. PMID 21850522
- [Background] Hamann J, Langer B, Winkler V, Busch R, Cohen R, Leucht S, Kissling W. Shared decision making for in-patients with schizophrenia. Acta Psychiatr Scand. 2006 Oct;114(4):265-73. doi: 10.1111/j.1600-0447.2006.00798.x. PMID 16968364
- [Background] Hamann J, Cohen R, Leucht S, Busch R, Kissling W. Do patients with schizophrenia wish to be involved in decisions about their medical treatment? Am J Psychiatry. 2005 Dec;162(12):2382-4. doi: 10.1176/appi.ajp.162.12.2382. PMID 16330606
- [Background] Joosten EA, DeFuentes-Merillas L, de Weert GH, Sensky T, van der Staak CP, de Jong CA. Systematic review of the effects of shared decision-making on patient satisfaction, treatment adherence and health status. Psychother Psychosom. 2008;77(4):219-26. doi: 10.1159/000126073. Epub 2008 Apr 16. PMID 18418028
- [Background] Malm U, Ivarsson B, Allebeck P, Falloon IR. Integrated care in schizophrenia: a 2-year randomized controlled study of two community-based treatment programs. Acta Psychiatr Scand. 2003 Jun;107(6):415-23. doi: 10.1034/j.1600-0447.2003.00085.x. PMID 12752017
- [Background] Malm UI, Ivarsson BA, Allebeck P. Durability of the efficacy of integrated care in schizophrenia: a five-year randomized controlled study. Psychiatr Serv. 2014 Aug 1;65(8):1054-7. doi: 10.1176/appi.ps.201300164. PMID 24932858
- [Background] Ekman I, Wolf A, Olsson LE, Taft C, Dudas K, Schaufelberger M, Swedberg K. Effects of person-centred care in patients with chronic heart failure: the PCC-HF study. Eur Heart J. 2012 May;33(9):1112-9. doi: 10.1093/eurheartj/ehr306. Epub 2011 Sep 15. PMID 21926072
- [Background] Olsson LE, Karlsson J, Ekman I. Effects of nursing interventions within an integrated care pathway for patients with hip fracture. J Adv Nurs. 2007 Apr;58(2):116-25. doi: 10.1111/j.1365-2648.2007.04209.x. PMID 17445014
- [Background] Chenoweth L, Forbes I, Fleming R, King MT, Stein-Parbury J, Luscombe G, Kenny P, Jeon YH, Haas M, Brodaty H. PerCEN: a cluster randomized controlled trial of person-centered residential care and environment for people with dementia. Int Psychogeriatr. 2014 Jul;26(7):1147-60. doi: 10.1017/S1041610214000398. Epub 2014 Mar 26. PMID 24666667
- [Background] Brownie S, Nancarrow S. Effects of person-centered care on residents and staff in aged-care facilities: a systematic review. Clin Interv Aging. 2013;8:1-10. doi: 10.2147/CIA.S38589. Epub 2013 Jan 3. PMID 23319855
- [Background] Rogers ES, Ralph RO, Salzer MS. Validating the empowerment scale with a multisite sample of consumers of mental health services. Psychiatr Serv. 2010 Sep;61(9):933-6. doi: 10.1176/ps.2010.61.9.933. PMID 20810594
- [Background] Ahlfors UG, Lewander T, Lindstrom E, Malt UF, Lublin H, Malm U. Assessment of patient satisfaction with psychiatric care. Development and clinical evaluation of a brief consumer satisfaction rating scale (UKU-ConSat). Nord J Psychiatry. 2001;55 Suppl 44:71-90. doi: 10.1080/080394801317084437. PMID 11860667
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Kinter ET, Schmeding A, Rudolph I, dosReis S, Bridges JF. Identifying patient-relevant endpoints among individuals with schizophrenia: an application of patient-centered health technology assessment. Int J Technol Assess Health Care. 2009 Jan;25(1):35-41. doi: 10.1017/S0266462309090059. PMID 19126249
- [Background] Nolte, Ellen, and Martin McKee, eds. Caring for people with chronic conditions: a health system perspective. McGraw-Hill Education (UK), 2008.
- [Background] Ashburner C, Meyer J, Johnson B, Smith C. Using action research to address loss of personhood in a continuing care setting. Illness, Crisis & Loss. 2004;12(1):23-37.
- [Background] Opler MG, Yang LH, Caleo S, Alberti P. Statistical validation of the criteria for symptom remission in schizophrenia: preliminary findings. BMC Psychiatry. 2007 Jul 24;7:35. doi: 10.1186/1471-244X-7-35. PMID 17650312
- [Background] Endicott J, Spitzer RL, Fleiss JL, Cohen J. The global assessment scale. A procedure for measuring overall severity of psychiatric disturbance. Arch Gen Psychiatry. 1976 Jun;33(6):766-71. doi: 10.1001/archpsyc.1976.01770060086012. PMID 938196
- [Background] Krippendorff, Klaus. Content analysis: An introduction to its methodology. Sage, 2004.
- [Background] Braun, Virginia, and Victoria Clarke.
- [Derived] Goulding A, Wiktorsson S, Allerby K, Ali L, Waern M. Service User and Next-of-Kin Experiences of Psychosis Inpatient Care After a Person-Centred Care Intervention. Issues Ment Health Nurs. 2025 Feb;46(2):138-147. doi: 10.1080/01612840.2024.2437429. Epub 2025 Jan 6. PMID 39761213
- [Derived] Allerby K, Gremyr A, Ali L, Waern M, Goulding A. Increasing person-centeredness in psychosis inpatient care: care consumption before and after a person-centered care intervention. Nord J Psychiatry. 2023 Aug;77(6):600-607. doi: 10.1080/08039488.2023.2199726. Epub 2023 Apr 21. PMID 37083029
- [Derived] Allerby K, Goulding A, Ali L, Waern M. Increasing person-centeredness in psychosis inpatient care: staff experiences from the Person-Centered Psychosis Care (PCPC) project. BMC Health Serv Res. 2022 May 3;22(1):596. doi: 10.1186/s12913-022-08008-z. PMID 35505358
- [Derived] Allerby K, Goulding A, Ali L, Waern M. Striving for a more person-centered psychosis care: results of a hospital-based multi-professional educational intervention. BMC Psychiatry. 2020 Nov 4;20(1):523. doi: 10.1186/s12888-020-02871-y. PMID 33148190
- [Derived] Goulding A, Allerby K, Ali L, Gremyr A, Waern M. Study protocol design and evaluation of a hospital-based multi-professional educational intervention: Person-Centred Psychosis Care (PCPC). BMC Psychiatry. 2018 Aug 30;18(1):269. doi: 10.1186/s12888-018-1852-2. PMID 30165822